CLINICAL TRIAL: NCT01168648
Title: Yoga for Stress Management in Health Care Personnel and Its Relation to the Hypothalamus-pituitary-adrenal(HPA)Axis
Brief Title: Yoga for Stress Management in Health Care Personnel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Ekhaga Foundation Stockholm Sweden (Unknown); Region Stockholm (Other Government)
Responsible Party: Astrid Grensman, MD, Karolinska Institutet, Center for Family and Community Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Ekhagastiftelsen 2001-5
Record Dates: First submitted 2010-07-22; First posted 2010-07-23 (Estimated); Last update posted 2010-07-23 (Estimated); Status verified 2010-07

CONDITIONS: Yoga; Stress, Psychological; Stress, Physiological
Keywords: Yoga; Stress; Stress management; Hypothalamus-pituitary-adrenal axis
MeSH Terms: conditions — Stress, Psychological | interventions — Yoga; Movement; Breathing Exercises; Meditation; RE1-silencing transcription factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Yoga as stress management (Experimental): The intervention consists of following a program of yoga at least three times a week for three months. The yoga program has been designed to reduce stress.
  Interventions: Behavioral: Yoga as stress management
- Control group (Active Comparator): The group rests without using any specific program for relaxation at least three times a week for three months.
  Interventions: Other: Rest without using any relaxation technique
- Yoga as stress management fewer tests (Other): Eight persons participated in the same intervention as the experimental arm but did not undergo the full range of tests because they did not meet all the inclusion criteria for the study, most commonly because of medication use or body mass index.
  Interventions: Behavioral: Yoga as stress management

INTERVENTIONS:
Behavioral: Yoga as stress management — Yoga specially designed to reduce stress is practiced for approximately 30 minutes at least three times a week for three months, once in a group session led by a trained yoga instructor and twice or more at home. The yoga techniques used are physical postures or movements, meditation and breathing exercises. Every time they do the techniques, participants fill in a form detailing how they feel before and after and providing information on the experience of doing the exercises.
  Other Names: Asanas(physical postures or movements); Pranayama (breathing exercises); Meditation
  Arms: Yoga as stress management; Yoga as stress management fewer tests
Other: Rest without using any relaxation technique — The participants rest at home at least 30 minutes, at least three times a week for three months and without using any relaxation technique
  Arms: Control group

SUMMARY:
The purpose of this study is to investigate if yoga can be an effective stress management technique for health care personnel.

DETAILED DESCRIPTION:
Stress, both job related and personal, is an increasing problem in the health care sector. Yoga is said to have a good stress-reducing effect.

The participants will provide blood, urine, and saliva samples. They will take part in two different stress tests. They will also fill in various qualitative questionnaires, including the Swedish questionnaire on health related quality of life (SWEDQUAL), Antonovsky's sense of coherence scale (KASAM), and the Job stress survey (JSS), both before the study starts and after 3 months of participation.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18-30
* healthy
* work in the health care sector

Exclusion Criteria:

* medication, including contraceptives and all medications or topical skin preparations with cortisone in any form (exception: hormone replacement therapy for hypothyroidism were included if their hormone levels were within the normal range)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2003-08; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Reduced cortisol secretion | Three months

SECONDARY OUTCOMES:
Reduced stress measured by qualitative questionnaires (SWEQUAL, JSS, KASAM) | Three months

CONTACTS AND LOCATIONS:
Overall Officials: Astrid M Grensman, MD, Principal Investigator — KI, Center for Family and Community Medicine; Bikash D Acharya, M sc in Psy, Principal Investigator — KI, Center for Family and Community Medicine
Locations (1):
- Center for Family and Community Medicine, KI, Huddinge, Stockholm County, Sweden